CLINICAL TRIAL: NCT00786422
Title: The EINSTEIN CYP Cohort Study Oral Direct Factor Xa Inhibitor Rivaroxaban in Patients With Acute Symptomatic Deep-vein Thrombosis or Pulmonary Embolism Using a Strong CYP 3A4 Inducer
Brief Title: Deep Vein Thrombosis Treatment With the Oral Direct Factor Xa Inhibitor Rivaroxaban in Patients Using a Strong CYP 3A4 Inducer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13238; 2008-003303-31 (EudraCT Number)
Record Dates: First submitted 2008-11-05; First posted 2008-11-06 (Estimated); Results first posted 2014-06-13 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-10

CONDITIONS: Venous Thrombosis; Deep Vein Thrombosis
Keywords: Embolism and Thrombosis; Pulmonary Embolism; Embolism; Venous Thrombosis; Thrombosis; Enzyme Inducers; CYP Inducers; Cohort Study; Pharmacologic Actions; Respiratory Tract Diseases; Lung Diseases; Vascular Diseases; Human Immunodeficiency Virus (HIV); Neurologic disease; Additional relevant MeSH terms:; Fibrin Modulating Agents; Anticoagulants; Therapeutic Uses; Hematologic Agents; Enzyme Inhibitors; Cardiovascular Diseases; Cardiovascular Agents
MeSH Terms: conditions — Venous Thrombosis; Embolism and Thrombosis; Pulmonary Embolism; Embolism; Thrombosis; Respiratory Tract Diseases; Lung Diseases; Vascular Diseases; Acquired Immunodeficiency Syndrome; Cardiovascular Diseases | interventions — Rivaroxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Rivaroxaban (Xarelto, BAY59-7939) (Experimental)
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939)

INTERVENTIONS:
Drug: Rivaroxaban (Xarelto, BAY59-7939) — Participants received 30 mg rivaroxaban bid (twice-daily) orally for the first 3 weeks followed by 20 mg rivaroxaban bid for the remainder of the 3-month treatment period.

SUMMARY:
This is a multicenter, cohort study evaluating an adapted rivaroxaban dose regimen in patients with acute, proximal deep-vein thrombosis (DVT) or acute pulmonary embolism (PE) who concomitantly use a strong cytochrome P450 isoenzyme 3A4 (CYP 3A4) inducer for the entire 3-month study duration.

DETAILED DESCRIPTION:
The following laboratory variables were determined at baseline at the local laboratories: Hemoglobin, platelets, activated partial thromboplastin time (aPTT), international normalized ratio (INR), alanine aminotransferase (ALT), and creatinine.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed acute symptomatic proximal deep- vein thrombosis and/or pulmonary embolism
* Concomitant use of a strong CYP 3A4 inducer, (i.e., carbamazepine, phenytoin, rifampicin/rifampin, and rifabutin)

Exclusion Criteria:

* Legal lower age limitations (country specific)
* Thrombectomy, insertion of a caval filter, or use of a fibrinolytic agent to treat the current episode of deep -vein thrombosis and/or pulmonary embolism
* Other indication for vitamin K antagonist (VKA) than deep -vein thrombosis and/or pulmonary embolism
* Concomitant use of strong CYP3A4 inhibitors (e.g., HIV protease inhibitors, systemic ketoconazole)
* Use of the strong CYP 3A4 inducers phenobarbital/primidone or St John's Wort

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2009-05; Primary Completion 2011-05 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (14):
- Redcliffe, Queensland, Australia
- Vienna, Vienna, Austria
- São Paulo, São Paulo, Brazil
- München, Bavaria, Germany
- Debrecen, Hungary
- Israel (2):
  - Ashkelon
  - Holon
- Pavia, Italy
- Amsterdam, Netherlands
- South Africa (5):
  - Johannesburg, Gauteng
  - Pretoria, Gauteng
  - Roodepoort, Gauteng
  - Somerset West, Western Cape
  - Worcester, Western Cape

REFERENCES:
- See also: Click here and search for information of Bayer products for Europe — http://www.clinicaltrialsregister.eu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with confirmed acute proximal symptomatic deep vein thrombosis (DVT) or acute pulmonary embolism (PE) were recruited at specialized study sites.
Pre-assignment Details: Out of 25 participants screened, 25 participants were assigned to treatment.
Period: Rivaroxaban Treatment
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939)
Started | 25
Completed | 14
Not Completed | 11
Not completed — Death | 2
Not completed — Final visit earlier than planned | 3
Not completed — Lack of Efficacy | 1
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 1
Not completed — Non-compliance with study drug treatment | 1
Not completed — Adverse Event | 2
Period: Follow-up Period
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939)
Started | 20 (Participants entered follow-up period. No reason documents for those not entering this period)
Completed | 17
Not Completed | 3
Not completed — Death | 1
Not completed — End-of-study done up to 4 days early | 2

BASELINE CHARACTERISTICS:
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939)
Number analyzed (Participants) | 25
Age, Customized [Number; unit: Participants]
  < 65 years | 23
  65 - 75 years | 1
  > 75 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 12
Race [Number; unit: Participants]
  White | 1
  Black | 23
  Other (mixed South African descent) | 1
Creatinine clearance [Number; unit: Participants] — Volume of blood plasma cleared of creatinine per time unit
  Participants
    <30 mL/min | 0
    30 - <50 mL/min | 0
    50 - <80 mL/min | 4
    > 80 mL/min | 21
Region of recruitment [Number; unit: Participants]
  South Africa - Yes | 25
  South Africa - No | 0
Participants with history of tuberculosis [Number; unit: Participants]
  History of tuberculosis | 20
  No history of tuberculosis | 5

OUTCOME MEASURES:

1. Primary Outcome: Pharmacodynamics - Prothrombin Time (PT), Baseline Value
Description: Prothrombin time (PT) is a global clotting test assessing the extrinsic pathway of the blood coagulation cascade. The test is sensitive for deficiencies of Factors II, V, VII, and X, with sensitivity being best for Factors V, VII, and X and less pronounced for Factor II. The initial read-out is in seconds. Mean and standard deviation (SD) values are presented for PT baseline.
Time Frame: The baseline value of prothrombin time is measured or calculated at a rivaroxaban concentration of 0 µg/L and is based on the observations that were made during the 3 months treatment period
Population: The pharmacokinetics/pharmacodynamics (PK/PD) population included all participants who received at least 1 dose of rivaroxaban and had at least 1 valid PK/PD sample after first administration
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939)
Number analyzed (Participants) | 19
Seconds | 15.8 (1.49)

2. Primary Outcome: Pharmacodynamics - Prothrombin Time (PT), Slope
Description: Prothrombin time (PT) is a global clotting test assessing the extrinsic pathway of the blood coagulation cascade. The test is sensitive for deficiencies of Factors II, V, VII, and X, with sensitivity being best for Factors V, VII, and X and less pronounced for Factor II. The initial read-out of PT is in seconds. The PT slope describes the linear increase of PT for one unit increase in concentration, thus the unit of PT slope is s*(µg/L)^-1. The final population PK/PD model included a fixed slope that was fitted to the data of the 19 patients that were eligible for evaluation. The estimated mean value (fixed/ the same for all patients in this study) is presented for PT slope.
Time Frame: Up to 3 months treatment
Population: as for outcome 1
Measure: Number; unit: s*(µg/L)^-1
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939)
Number analyzed (Participants) | 19
s*(µg/L)^-1 | 0.0389 (NA)

3. Primary Outcome: Pharmacokinetics - AUC(0-24)ss (Area Under the Measurement Versus Time Curve From Time 0 to 24 Hours After First Dosing on a Day at Steady State) of Rivaroxaban
Description: AUC(0-24)ss was predicted from rivaroxaban plasma concentrations for each individual participant and was only considered for the time period during which participants concomitantly received rivaroxaban and a strong cytochrome P450 isoenzyme 3A4 (CYP3A4) inducer.
Time Frame: 0 (predose), 1, 2, 3, 4, 6, 8, 12, and 24 h after first administration of rivaroxaban
Population: as for outcome 1
Measure: Median (90% Confidence Interval); unit: (µg*h)/L
Groups:
- Rivaroxaban Initial Treatment: Participants received 30 mg rivaroxaban bid (twice-daily) orally for the first 3 weeks.
- Rivaroxaban Extended Treatment: Participants received 20 mg rivaroxaban bid (twice-daily) orally for the remainder of the 3-month treatment period.
Arm/Group | Rivaroxaban Initial Treatment | Rivaroxaban Extended Treatment
Number analyzed (Participants) | 19 | 18
(µg*h)/L | 2836 [1259 to 6877] | 2319 [1059 to 5782]

4. Primary Outcome: Pharmacokinetics - Cmax,ss (Maximum Observed Drug Concentration in Measured Matrix at Steady State During a Dosage Interval) of Rivaroxaban
Description: Cmax,ss was predicted from rivaroxaban plasma concentrations for each individual participant and was only considered for the time period during which participants concomitantly received rivaroxaban and a strong CYP3A4 inducer.
Time Frame: 0 (predose), 1, 2, 3, 4, 6, 8, 12, and 24 h after first administration of rivaroxaban
Population: as for outcome 1
Measure: Median (90% Confidence Interval); unit: µg/L
Arm/Group | Rivaroxaban Initial Treatment | Rivaroxaban Extended Treatment
Number analyzed (Participants) | 19 | 18
µg/L | 200 [150 to 386] | 167 [126 to 324]

5. Primary Outcome: Pharmacokinetics - Cmin,ss (Minimum Observed Drug Concentration in Measured Matrix at Steady State During a Dosage Interval) of Rivaroxaban
Description: Cmin,ss was predicted for each individual participant from rivaroxaban plasma concentrations and was only considered for the time period during which participants concomitantly received rivaroxaban and a strong CYP3A4 inducer.
Time Frame: 0 (predose), 1, 2, 3, 4, 6, 8, 12, and 24 h after first administration of rivaroxaban
Population: as for outcome 1
Measure: Median (90% Confidence Interval); unit: µg/L
Arm/Group | Rivaroxaban Initial Treatment | Rivaroxaban Extended Treatment
Number analyzed (Participants) | 19 | 18
µg/L | 42 [1 to 170] | 35 [1 to 143]

6. Primary Outcome: Percentage of Participants With Clinically Relevant Bleeding (i.e. Major Bleeding and Clinically Relevant Non-major Bleeding)
Description: All events were adjudicated and confirmed by a central independent adjudication committee. Clinically relevant bleeding included major bleeding (overt bleeding associated with 2 g/dL or greater fall in hemoglobin, leading to a transfusion of 2 or more units of packed red blood cells or whole blood, occurring in a critical site or contributing to death) and non-major bleeding associated with medical intervention, unscheduled physician contact, (temporary) cessation of study treatment, discomfort for the participants such as pain, or impairment of activities of daily life.
Time Frame: Up to 3 months treatment and during subsequent 2 days
Population: The safety population consisted of all participants who received at least 1 dose of rivaroxaban.
Measure: Number; unit: Percentage of participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939)
Number analyzed (Participants) | 25
Percentage of participants
  Any confirmed bleeding | 12.0
  Clinically relevant non-major bleeding | 8.0
  Trivial bleeding | 8.0

7. Secondary Outcome: Percentage of Participants With Symptomatic Recurrent Venous Thromboembolism [VTE] (i.e. the Composite of Recurrent Deep Vein Thrombosis [DVT] or Non-fatal or Fatal Pulmonary Embolism [PE]) Until the Intended End of Study Treatment
Description: All events were adjudicated and confirmed by a central independent adjudication committee. The composite efficacy outcome symptomatic recurrent VTE was analyzed descriptively, with the components: Death due to PE, death for which PE cannot be excluded, symptomatic PE and DVT, symptomatic recurrent PE only, and symptomatic recurrent DVT only up to the end of intended treatment period (3 months; 98 study days) and on-treatment (up to 2 days after stop of study drug).
Time Frame: Up to 3 months treatment and during subsequent 30-day observational period for an individual participant
Population: The safety population consisted of all participants who received at least 1 dose of rivaroxaban.
Measure: Number; unit: Percentage of participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939)
Number analyzed (Participants) | 25
Percentage of participants
  symptomatic recurrent VTE (composite) | 8.0
  Death | 4.0
  Symptomatic recurrent deep vein thrombosis only | 4.0

8. Secondary Outcome: Percentage of Participants With All Deaths
Description: All deaths were adjudicated by a central independent adjudication committee. Participants who died for any reason were counted for this measure.
Time Frame: Up to 3 months and on-treatment (up to 2 days after stop of study drug) plus an observational period planned for one month
Population: All participants
Measure: Number; unit: Percentage of participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939)
Number analyzed (Participants) | 25
Percentage of participants | 12.0

9. Secondary Outcome: Percentage of Participants With Treatment Emergent Deaths - 7 Days Window
Description: Treatment emergent deaths were adjudicated by a central independent adjudication committee. Participants who died from treatment emergent adverse events were counted for this measure.
Time Frame: Up to 3 months treatment and during subsequent 7 days
Population: All participants
Measure: Number; unit: Percentage of participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939)
Number analyzed (Participants) | 25
Percentage of participants | 8.0

10. Secondary Outcome: Percentage of Participants With Other Vascular Events
Description: All events were adjudicated and confirmed by a central independent adjudication committee. Other vascular events comprised ST segment elevation myocardial infarction (STEMI), non-ST segment elevation myocardial infarction (NSTEMI), unstable angina (UA), ischemic stroke, transient ischemic attack (TIA), non-central nervous system systemic embolism and vascular death.
Time Frame: Up to 3 months treatment and during subsequent 1 day
Population: The safety population consisted of all participants who received at least 1 dose of rivaroxaban.
Measure: Number; unit: Percentage of participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939)
Number analyzed (Participants) | 25
Percentage of participants | 0.0

ADVERSE EVENTS:
Time Frame: For the whole study, adverse event (AE) data were collected during the study course of 25 months. For the individual patient, AE were collected during a treatment period planned for three months plus an observational period planned for one month.
Description: Abbreviations used:Human Immunodeficiency Virus (HIV)
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939)
Serious Adverse Events (participants affected / at risk) | 5/25
Other Adverse Events (participants affected / at risk) | 14/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rivaroxaban (Xarelto, BAY59-7939) (N=25)
Death (General disorders) | 2
Sudden death (General disorders) | 1
Hepatitis (Hepatobiliary disorders) | 1
Meningitis cryptococcal (Infections and infestations) | 1
Vascular dementia (Nervous system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rivaroxaban (Xarelto, BAY59-7939) (N=25)
Neutropenia (Blood and lymphatic system disorders) | 1
Tachycardia (Cardiac disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Oedema (General disorders) | 1
Oedema peripheral (General disorders) | 1
Cellulitis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 3
HIV test positive (Investigations) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Haematoma (Vascular disorders) | 1
Vein pain (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator, whilst free to utilize data derived from the study for scientific purposes, must discuss any publication with Bayer prior to release and obtain written consent of Bayer on the intended publication. The investigator must send a draft manuscript of the publication or abstract to Bayer thirty days in advance of submission in order to obtain approval prior to submission of the final version for publication.